CLINICAL TRIAL: NCT02520427
Title: A Phase 1 First-in-human Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of AMG 330 Administered as Continuous Intravenous Infusion in Subjects With Myeloid Malignancies
Brief Title: A Phase 1 Study of AMG 330 in Subjects With Myeloid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Amgen strategic business decision to cancel following portfolio review, re-prioritization.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20120252; 2014-004462-20 (EudraCT Number)
Record Dates: First submitted 2015-06-17; First posted 2015-08-11 (Estimated); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-02

CONDITIONS: Relapsed/Refractory AML; Minimal Residual Disease Positive AML; Myelodysplastic Syndrome
Keywords: Amgen; Phase 1; Clinical Trial; Oncology/Hematology; Relapsed/Refractory AML; Immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Neoplasms | interventions — AMG 330

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1: Relapsed/Refractory Acute Myeloid Leukemia (R/R AML) (Experimental)
  Interventions: Drug: AMG 330
- Group 2: Minimal Residual Disease Positive (MRD+) AML (Experimental)
  Interventions: Drug: AMG 330
- Group 3: Myelodysplastic syndrome (MDS) (Experimental)
  Interventions: Drug: AMG 330
- Group 4: R/R AML with alternative pretreatment (Experimental)
  Interventions: Drug: AMG 330
- Group 5: R/R AML with alternative dose schedule (Experimental)
  Interventions: Drug: AMG 330

INTERVENTIONS:
Drug: AMG 330 — 0.5 µg/day - 1.6 mg/day cIV infusion administered in cycles from 14 to 28 days.

SUMMARY:
The purpose of this First-in-Human Phase 1 study is to determine if AMG 330 given as a continuous IV infusion is safe and tolerable in adult subjects that have myeloid malignancies, and to determine the maximum tolerated dose and/or a biologically active dose. The study will be conducted in multiple sites and test increasing doses of AMG 330. The safety of subjects will be monitored by intensive assessment of vital signs, electrocardiograms, physical examinations, and laboratory tests.

ELIGIBILITY:
Inclusion criteria:

* Informed consent provided
* 18 years or older
* Relapsed/refractory AML: AML as defined by the WHO Classification persisting or recurring following one or more treatment courses except promyelocytic leukemia (APML)

Exclusion criteria:

* Active extramedullary AML in testes or central nervous system (CNS)
* Known hypersensitivity to immunoglobulins or to any other component of the IP formulation (eg, sucrose, captisol, potassium, polysorbate 80, citrate, lysine)
* Prior malignancy (other than in situ cancer) unless treated with curative intent and without evidence of disease for > 1 years before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2022-01-09 (Actual); Study Completion 2022-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Research Site, Duarte, California
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Germany (3):
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Klinikum der Universität München Campus Grosshadern, München
  - Universitatsklinikum Ulm, Ulm
- Netherlands (2):
  - Research Site, Amsterdam
  - Erasmus Medisch Centrum, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 9 research centers in the United States, Germany and the Netherlands and participated in the trial from August 2015 to December 2021.
Pre-assignment Details: 95 participants were enrolled and received treatment.
Groups:
- Group 1 - Cohort 1 AMG 330 0.5 µg/Day: Participants with R/R AML (Group 1) received AMG 330 0.5 µg/day as a 14 day continuous infusion (cIV).
- Group 1 - Cohort 2 AMG 330 1.5 µg/Day: Participants with R/R AML (Group 1) received AMG 330 1.5 µg/day as a 14 day cIV.
- Group 1 - Cohort 3 AMG 330 4 µg/Day: Participants with R/R AML (Group 1) received AMG 330 4 µg/day as a 14 day cIV.
- Group 1 - Cohort 4 AMG 330 10 µg/Day: Participants with R/R AML (Group 1) received AMG 330 10 µg/day as a 14 day cIV.
- Group 1 - Cohort 5 AMG 330 30 µg/Day: Participants with R/R AML (Group 1) received AMG 330 30 µg/day as a 14 day cIV.
- Group 1 - Cohort 6 AMG 330 10/30 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at an initial step dose of 10 µg/day and then the target dose of 30 µg/day as a 14 day cIV.
- Group 1 - Cohort 7 AMG 330 10/60 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at an initial step dose of 10 µg/day and then the target dose of 60 µg/day as a 14 day cIV.
- Group 1 - Cohort 8 AMG 330 10/120 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at an initial step dose of 10 µg/day and then the target dose of 120 µg/day as a 14 day cIV.
- Group 1 - Cohort 9 AMG 330 10/240 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at an initial step dose of 10 µg/day and then the target dose of 240 µg/day as a 14 day cIV.
- Group 1 - Cohort 10 AMG 330 10/480 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at an initial step dose of 10 µg/day and then the target dose of 480 µg/day as a 14 day cIV.
- Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at an initial daily step dose of 10 µg/day and a second step dose of 60 µg/day, and then the target dose of 240 µg/day as a 28 day cIV.
- Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day: Participants with R/R AML (Group 1) received AMG 330 at an initial daily step dose of 10 µg/day and a second step dose of 60 µg/day, then the target dose of 240 µg/day as a 28 day cIV.
- Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at an initial daily step dose of 10 µg/day and a second step dose of 60 µg/day, and then the target dose of 360 µg/day as a 28 day cIV.
- Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at an initial daily step dose of 10 µg/day and a second step dose of 60 µg/day, and then the target dose of 480 µg/day as a 28 day cIV.
- Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at an initial daily step dose of 10 µg/day and a second step dose of 240 µg/day, and then the target dose of 600 µg/day as a 28 day cIV.
- Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at initial daily step doses of 10, 240 and 600 µg/day and then the target dose of 720 µg/day as a 28 day cIV.
- Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at initial daily step doses of 10, 240 and 600 µg/day and then the target dose of 840 µg/day as a 28 day cIV.
- Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at initial daily step doses of 10, 240 and 600 µg/day and then the target dose of 960 µg/day as a 28 day cIV.
- Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at initial daily step doses of 10, 240, 600, and 960 µg/day and then the target dose of 1300 µg/day as a 28 day cIV.
- Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day: Participants with R/R AML (Group 1) received AMG 330 at initial daily step doses of 10, 60, 240, 600, and 960 µg/day and then the target dose of 1600 µg/day as a 28 day cIV.
- Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day: Participants with MRD+ AML (Group 2) received AMG 330 at initial daily step doses of 30 µg/day for up to 2 days, 240 µg/day for up to 5 days and then the target dose of 600 µg/day as a 28 day cIV.
- Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day: Participants with MRD+ AML (Group 2) received AMG 330 at initial step daily doses of 30 µg/day for up to 2 days, 240 µg/day for up to 5 days and then the target dose of 840 µg/day as a 28 day cIV.
- Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day: Participants with MDS (Group 3) received AMG 330 at initial daily step doses of 30 µg/day for up to 2 days and 240 µg/day for up to 5 days and then the target dose of 600 µg/day for a total of a 28 day cIV.
- Group 4 - Etanercept and AMG 330: Participants with R/R AML received etanercept 50 mg as a subcutaneous (SC) injection in combination with AMG 330. Participants received AMG 330 at initial daily step doses of 10 µg/day for 2 days, 60 µg/day for 3 days and 240 µg/day for 9 days for a total of a 14 day cIV.
  Participants received etanercept 1 day before first AMG 330 administration and on Day 4 of each cycle.
- Group 4 - Etanercept, Dexamethasone and AMG 330: Participants with R/R AML received etanercept 50 mg as a SC injection and dexamethsone 8 mg IV infusion in combination with AMG 330. Participants received AMG 330 at initial daily step doses of 10 µg/day for 2 days, 60 µg/day for 3 days and 240 µg/day for 9 days for a total of a 14 day cIV.
  Participants received etanercept 1 day before first AMG 330 administration and on Day 4 of each cycle.
  Participants received dexamethasone 1 hour before AMG 330 dose.
- Group 4: Tocilizumab, Dexamethasone and AMG 330: Participants with R/R AML received tocilizumab 8 mg/kg IV infusion and dexamethsone 8 mg IV infusion in combination with AMG 330. Participants received AMG 330 at initial daily step doses of 10 µg/day for 2 days, 60 µg/day for 3 days and 240 µg/day for 9 days for a total of a 14 day cIV.
  Participants received tocilizumab on Day 1, 1 hour before the 1st dose of AMG 330 of each cycle.
  Participants received dexamethasone 1 hour before AMG 330 dose.
Period: Overall Study
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330
Started | 1 | 1 | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 4 | 7 | 3 | 3 | 6 | 3 | 5 | 4 | 5 | 8 | 4 | 2 | 4 | 3 | 4 | 1
Completed | 0 | 1 | 2 | 3 | 3 | 3 | 4 | 4 | 3 | 2 | 4 | 7 | 2 | 2 | 5 | 3 | 2 | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 1
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 3 | 5 | 2 | 0 | 1 | 0 | 1 | 0
Not completed — Decision by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 2 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330 | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 4 | 7 | 3 | 3 | 6 | 3 | 5 | 4 | 5 | 8 | 4 | 2 | 4 | 3 | 4 | 1 | 95
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 0 | 1 | 2 | 2 | 1 | 2 | 3 | 1 | 2 | 2 | 2 | 5 | 3 | 2 | 4 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2 | 2 | 3 | 0 | 58
  65-74 years | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 3 | 2 | 0 | 2 | 1 | 1 | 0 | 31
  75-84 years | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 3 | 2 | 2 | 3 | 2 | 1 | 2 | 1 | 3 | 2 | 2 | 3 | 1 | 1 | 1 | 2 | 3 | 0 | 42
  Male | 0 | 0 | 2 | 1 | 1 | 3 | 3 | 4 | 1 | 1 | 2 | 4 | 1 | 2 | 4 | 2 | 2 | 2 | 3 | 5 | 3 | 1 | 3 | 1 | 1 | 1 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 16
  Not Hispanic or Latino | 1 | 1 | 3 | 3 | 3 | 1 | 3 | 4 | 4 | 2 | 2 | 6 | 3 | 3 | 5 | 3 | 4 | 3 | 4 | 8 | 4 | 1 | 3 | 2 | 2 | 1 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  Asian | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 16
  Black (or African American) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 0 | 1 | 3 | 1 | 2 | 1 | 4 | 4 | 3 | 3 | 3 | 7 | 2 | 1 | 5 | 2 | 4 | 2 | 4 | 6 | 2 | 1 | 3 | 2 | 2 | 1 | 69
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT)
Description: A participant was not DLT-evaluable if they dropped out before completion of the DLT window (14 days) for reasons other than an adverse event related to study drug or the participant had not received investigational product (IP) treatment for at least 14 days at the target dose for a 3- or 4-week cycle or at least 7 days at a target dose for a 2- week cycle. Furthermore, following drug interruptions, if a participant was unable to complete 2 repeat cycles for reasons other than DLT, the participant was not DLT evaluable.
Time Frame: Day 1 to Day 14
Population: DLT-evaluable Analysis Set: All DLT-evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 5 | 3 | 2 | 3 | 2 | 4 | 0
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |

2. Secondary Outcome: Number of Participants Who Experienced an Incident of Anti-AMG 330 Antibody Formation
Description: Number of participants with a binding anti-body positive result at any timepoint post-baseline who had a negative or no result at baseline.
Time Frame: Baseline until the end of study, up to approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 4 | 7 | 3 | 3 | 6 | 3 | 5 | 4 | 5 | 7 | 4 | 2 | 4 | 3 | 4 | 1
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0

3. Secondary Outcome: Response Rate in Participants With R/R AML
Description: Response for participants with R/R AML was defined as the percentage of participants with complete response (CR)/complete remission with incomplete count recovery (CRi)/morphologic leukemia-free state (MLFS) [per modified international working group (IWG) criteria] or complete remission with partial hematologic recovery (CRh).
Time Frame: From first dose of IP (Day 1) until the end of study, up to approximately 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 4 | 7 | 3 | 3 | 6 | 3 | 5 | 4 | 5 | 8 | 3 | 4 | 1
Percentage of participants | 0.0 (0.0) [0.0 to 97.5] | 100.0 (2.5) [2.5 to 100.0] | 0.0 (0.0) [0.0 to 70.8] | 0.0 (0.0) [0.0 to 70.8] | 0.0 (0.0) [0.0 to 70.8] | 0.0 (0.0) [0.0 to 70.8] | 0.0 (0.0) [0.0 to 60.2] | 25.0 (0.6) [0.6 to 80.6] | 25.0 (0.6) [0.6 to 80.6] | 0.0 (0.0) [0.0 to 70.8] | 25.0 (0.6) [0.6 to 80.6] | 14.3 (0.4) [0.4 to 57.9] | 0.0 (0.0) [0.0 to 70.8] | 0.0 (0.0) [0.0 to 70.8] | 33.3 (4.3) [4.3 to 77.7] | 33.3 (0.8) [0.8 to 90.6] | 0.0 (0.0) [0.0 to 52.2] | 0.0 (0.0) [0.0 to 60.2] | 0.0 (0.0) [0.0 to 52.2] | 0.0 (0.0) [0.0 to 36.9] | 0.0 (0.0) [0.0 to 70.8] | 0.0 (0.0) [0.0 to 60.2] | 0.0 (0.0) [0.0 to 97.5]

4. Secondary Outcome: Response Rate in Participants With MRD-positive AML
Description: Response for participants with MRD-positive AML was defined as the percentage of participants with a conversion from MRD+ status with 0.1% threshold to CRMDR- or CRiMD-.
Time Frame: From first dose of IP (Day 1) until the end of study, up to approximately 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day
Number analyzed (Participants) | 4 | 2
Percentage of participants | 25.0 (0.6) [0.6 to 80.6] | 0.0 (0.0) [0.0 to 84.2]

5. Secondary Outcome: Response Rate in Participants With MDS
Description: Response for participants with MDS was defined as the percentage of participants with CR or marrow complete remission per IWG.
Time Frame: From first dose of IP (Day 1) until the end of study, up to approximately 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day
Number analyzed (Participants) | 4
Percentage of participants | 25.0 (0.6) [0.6 to 80.6]

6. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the interval from the date of the first disease assessment indicating an overall response to the first documented relapse, disease progression, or death due to any cause, whichever occurs first.
Time Frame: From first dose of IP (Day 1) until the end of study, up to approximately 6 months
Population: Per the Statistical Analysis Plan, duration of response was only planned to be measured in the expansion cohorts. Therefore, this endpoint was not summarized due to early termination of the trial prior to dose expansion.
Groups:
- Group 1: All participants with R/R AML who received AMG 330 at doses ranging from 0.5 µg/day to 1600 µg/day as either a 14 day or 28 day cIV.
- Group 2: All participants with MRD+ AML who received AMG 330 at doses ranging from 30 µg/day to 840 µg/day as a 28 day cIV.
- Group 3: All participants with MDS who received AMG 330 at doses ranging from 30 µg/day up to 600 µg/day as a 28 day cIV.
- Group 4: All participants with R/R AML who received either etanercept 50 mg SC injection or tocilizumab 8 mg/kg IV infusion with or without dexamethsone 8 mg IV infusion in combination with AMG 330.
  Doses of AMG 330 ranged from 10 µg/day to 240 µg/day as a 14 day cIV.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Time to Response
Description: Time to response was defined as the interval from the first administration of AMG 330 to the first documentation of response.
Time Frame: From first dose of IP (Day 1) until the end of study, up to approximately 6 months
Population: Per the Statistical Analysis Plan, time to response was only planned to be measured in the expansion cohorts. Therefore, this endpoint was not summarized due to early termination of the trial prior to dose expansion.
Groups:
- Group 3: All participants with MDS who received AMG 330 at doses ranging from 30 µg/day to 600 µg/day as a 28 day cIV.
- Group 4: All participants with R/R AML who received either etanercept 50 mg SC injection or tocilizumab mg/kg IV infusion with or without dexamethsone 8 mg IV infusion, in combination with AMG 330.
  Doses of AMG 330 ranged from 10 µg/day to 240 µg/day as a 14 day cIV.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Event-free Survival
Description: Event-free survival was defined as the interval from first administration of AMG 330 to the earliest of date of treatment failure, relapse for responders, or death due to any cause.
Time Frame: From first dose of IP (Day 1) until the end of study, up to approximately 6 months
Population: Per the Statistical Analysis Plan, event-free survival was only planned to be measured in the expansion cohorts. Therefore, this endpoint was not summarized due to early termination of the trial prior to dose expansion.
Groups:
- Group 4: All participants with R/R AML who received either etanercept 50 mg SC injection or tocilizumab mg/kg IV injection with or without dexamethsone 8 mg IV infusion, in combination with AMG 330.
  Doses of AMG 330 ranged from 10 µg/day to 240 µg/day as a 14 day cIV.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from enrollment until death due to any cause.
Time Frame: Baseline until the end of study, up to approximately 6 months
Population: Per the Statistical Analysis Plan, overall survival was only planned to be measured in the expansion cohorts. Therefore, this endpoint was not summarized due to early termination of the trial prior to dose expansion.
Groups:
- Group 2: All participants with MRD+ AML who received AMG 300 at doses ranging from 30 µg/day to 840 µg/day as a 28 day cIV.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: 14 Day Infusion Duration: Terminal Half Life (t1/2 z) of AMG 330
Time Frame: 14 day infusion duration: Pre-dose to 48 hours from the start of infusion, and days 4, 8, 11, 15, 16 and 22 of Cycle 1 for Group 1 and days 8, 15 and 16 for Group 4 (each cycle was 28 days)
Population: Includes all participants who had analyzable samples.
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 0 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0
hours |  |  | 2.68 (2.68) [2.68 to 2.68] | 3.28 (2.90) [2.90 to 4.48] |  | 4.03 (2.59) [2.59 to 4.30] | 5.34 (5.05) [5.05 to 5.62] | 8.07 (8.07) [8.07 to 8.07] | 7.34 (7.20) [7.20 to 7.49] |  |  |  |

11. Secondary Outcome: 28 Day Infusion Duration: t1/2 z of AMG 330
Time Frame: Pre-dose to 48 hours from the start of infusion, and days 8, 15, 22, 29, and 30 of Cycle 1 (each cycle was 36 days)
Population: Includes all participants who had analyzable samples.
Measure: Median (Full Range); unit: Hours
Arm/Group | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day
Number analyzed (Participants) | 1 | 1 | 0 | 2 | 3 | 1 | 3 | 2 | 3 | 2 | 1 | 2 | 3
Hours | 8.34 (8.34) [8.34 to 8.34] | 6.49 (6.49) [6.49 to 6.49] |  | 4.57 (4.47) [4.47 to 4.67] | 5.03 (4.37) [4.37 to 8.07] | 4.96 (4.96) [4.96 to 4.96] | 8.67 (7.71) [7.71 to 9.18] | 3.71 (3.21) [3.21 to 4.22] | 4.99 (2.58) [2.58 to 5.41] | 3.80 (2.90) [2.90 to 4.71] | 9.14 (9.14) [9.14 to 9.14] | 4.22 (3.32) [3.32 to 5.13] | 6.43 (6.30) [6.30 to 7.34]

12. Secondary Outcome: 14 Day Infusion Duration: Steady State Serum Concentration After End of Infusion (Css) of AMG 330
Time Frame: Pre-dose to 48 hours from the start of infusion, and days 4, 8, 11, 15, 16 and 22 of Cycle 1 for Group 1 and days 8, 15 and 16 for Group 4 (each cycle was 28 days)
Population: Includes all participants who had analyzable samples.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 2 | 0 | 1 | 0
ng/mL | 0.00 (0.00) [0.00 to 0.00] | 0.0231 (0.0231) [0.0231 to 0.0231] | 0.0541 (0.0378) [0.0378 to 0.0608] | 0.158 (0.0856) [0.0856 to 0.290] | 0.221 (0.220) [0.220 to 0.221] | 0.155 (0.134) [0.134 to 0.234] | 0.325 (0.240) [0.240 to 0.410] | 0.610 (0.390) [0.390 to 0.830] | 2.29 (1.16) [1.16 to 2.52] | 3.97 (2.97) [2.97 to 4.96] |  | 0.952 (0.952) [0.952 to 0.952] |

13. Secondary Outcome: 28 Day Infusion Duration: Css After End of Infusion of AMG 330
Time Frame: Pre-dose to 48 hours from the start of infusion, and days 8, 15, 22, 29, and 30 of Cycle 1 (each cycle was 36 days)
Population: Includes all participants who had analyzable samples.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330 | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day
Number analyzed (Participants) | 4 | 3 | 1 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 1 | 1 | 0 | 1 | 0 | 3
ng/mL | 0.440 (0.200) [0.200 to 5.13] | 1.83 (1.07) [1.07 to 2.02] | 1.56 (1.56) [1.56 to 1.56] | 5.92 (3.61) [3.61 to 8.23] | 5.95 (4.62) [4.62 to 19.5] | 7.36 (2.09) [2.09 to 12.6] | 3.20 (2.24) [2.24 to 4.16] | 24.2 (5.46) [5.46 to 63.0] | 7.52 (5.82) [5.82 to 13.6] | 1.79 (1.37) [1.37 to 2.21] | 8.40 (8.40) [8.40 to 8.40] | 1.14 (1.14) [1.14 to 1.14] |  | 0.952 (0.952) [0.952 to 0.952] |  | 1.76 (0.920) [0.920 to 2.00]

14. Secondary Outcome: 14 Day Infusion Duration: Volume of Distribution at Steady State (Vz) of AMG 330
Time Frame: as for outcome 12
Population: Includes all participants who had analyzable samples.
Measure: Median (Full Range); unit: Liters
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 0 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Liters |  |  | 11.9 (11.9) [11.9 to 11.9] | 17.0 (6.02) [6.02 to 23.0] |  | 31.0 (30.1) [30.1 to 57.9] | 62.7 (49.5) [49.5 to 76.0] | 149 (149) [149 to 149] | 44.1 (42.9) [42.9 to 45.4] |  |  |  |

15. Secondary Outcome: 28 Day Infusion Duration: Vz of AMG 330
Time Frame: Pre-dose to 48 hours from the start of infusion, and days 8, 15, 22, 29, and 30 of Cycle 1 (each cycle was 36 day)
Population: Includes all participants who had analyzable samples.
Measure: Median (Full Range); unit: Liters
Arm/Group | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day
Number analyzed (Participants) | 1 | 1 | 0 | 2 | 3 | 1 | 2 | 2 | 3 | 2 | 1 | 1 | 3
Liters | 293 (293) [293 to 293] | 69.6 (69.6) [69.6 to 69.6] |  | 33.1 (19.6) [19.6 to 46.7] | 47.1 (9.69) [9.69 to 58.7] | 19.8 (19.8) [19.8 to 19.8] | 165 (107) [107 to 223] | 8.79 (3.98) [3.98 to 13.6] | 63.8 (18.2) [18.2 to 89.4] | 76.6 (76.3) [76.3 to 76.8] | 54.9 (54.9) [54.9 to 54.9] | 105 (105) [105 to 105] | 60.2 (46.4) [46.4 to 98.8]

16. Secondary Outcome: 14 Day Infusion Duration: Clearance at Steady State (CL) for AMG 330
Time Frame: as for outcome 12
Population: Includes all participants who had analyzable samples.
Measure: Median (Full Range); unit: L/hr
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330
Number analyzed (Participants) | 0 | 1 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 2 | 0 | 1 | 0
L/hr |  | 2.71 (2.71) [2.71 to 2.71] | 3.08 (2.74) [2.74 to 4.41] | 2.64 (1.44) [1.44 to 4.87] | 5.67 (5.66) [5.66 to 5.68] | 8.06 (5.34) [5.34 to 9.33] | 8.26 (6.10) [6.10 to 10.4] | 9.42 (6.02) [6.02 to 12.8] | 4.37 (3.97) [3.97 to 8.62] | 5.38 (4.03) [4.03 to 6.73] |  | 10.5 (10.5) [10.5 to 10.5] |

17. Secondary Outcome: 28 Day Infusion Duration: CL of AMG 330
Time Frame: Pre-dose to 48 hours from the start of infusion, and days 8, 15, 22, 29, and 30 of Cycle 1 (each cycle was 36 days)
Measure: Median (Full Range); unit: L/hr
Arm/Group | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day
Number analyzed (Participants) | 4 | 3 | 1 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 1 | 1 | 3
L/hr | 22.8 (1.95) [1.95 to 50.0] | 8.20 (7.43) [7.43 to 14.0] | 12.8 (12.8) [12.8 to 12.8] | 4.98 (3.04) [3.04 to 6.93] | 5.04 (1.54) [1.54 to 6.49] | 9.76 (2.77) [2.77 to 16.7] | 13.7 (9.62) [9.62 to 17.9] | 2.23 (0.860) [0.860 to 9.92] | 8.87 (4.90) [4.90 to 11.5] | 14.8 (11.3) [11.3 to 18.2] | 4.17 (4.17) [4.17 to 4.17] | 21.9 (21.9) [21.9 to 21.9] | 5.68 (5.00) [5.00 to 10.9]

18. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: The severity of TEAEs were graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 criteria. The general guideline for assessment ranged from Grade 1 to 5, with higher grades indicating a worse outcome, and included: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, and Grade 5 = death.
Time Frame: Day 1 until 30 days after last dose. Median duration of treatment was: Group 1 - 29.0 days; Group 2 - 29.0 days; Group 3 - 49.50 days; Group 4 - 23.50 days
Population: Safety Analysis Set: All participants that were enrolled and received at least 1 dose of AMG 330.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 4 | 7 | 3 | 3 | 6 | 3 | 5 | 4 | 5 | 8 | 4 | 2 | 4 | 3 | 4 | 1
Participants
  All TEAEs | 1 | 1 | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 4 | 7 | 3 | 3 | 6 | 3 | 5 | 4 | 5 | 8 | 4 | 2 | 4 | 3 | 4 | 1
  Grade 1 | 1 | 1 | 2 | 3 | 2 | 3 | 4 | 4 | 4 | 3 | 4 | 7 | 3 | 3 | 6 | 3 | 5 | 4 | 5 | 7 | 4 | 2 | 4 | 3 | 4 | 1
  Grade 2 | 1 | 1 | 2 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 4 | 6 | 3 | 3 | 6 | 3 | 5 | 4 | 5 | 8 | 4 | 2 | 4 | 3 | 4 | 1
  Grade 3 | 1 | 1 | 2 | 3 | 3 | 3 | 4 | 4 | 2 | 3 | 4 | 6 | 3 | 2 | 5 | 3 | 4 | 3 | 5 | 8 | 3 | 2 | 4 | 3 | 3 | 1
  Grade 4 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 2 | 2 | 4 | 1 | 0 | 3 | 2 | 4 | 4 | 3 | 5 | 1 | 2 | 4 | 2 | 1 | 1
  Grade 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Mortality: Day 1 until end of study; median (min, max) time on study was 1.45 (0.26, 7.85) months. Adverse Events: Day 1 until 30 days after last dose. Median duration of treatment was: Group 1 - 29.0 days; Group 2 - 29.0 days; Group 3 - 49.50 days; Group 4 - 23.50 days
Description: Mortality is reported for all participants randomized.
  Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Group 1 - Cohort 1 AMG 330 0.5 µg/Day | Group 1 - Cohort 2 AMG 330 1.5 µg/Day | Group 1 - Cohort 3 AMG 330 4 µg/Day | Group 1 - Cohort 4 AMG 330 10 µg/Day | Group 1 - Cohort 5 AMG 330 30 µg/Day | Group 1 - Cohort 6 AMG 330 10/30 µg/Day | Group 1 - Cohort 7 AMG 330 10/60 µg/Day | Group 1 - Cohort 8 AMG 330 10/120 µg/Day | Group 1 - Cohort 9 AMG 330 10/240 µg/Day | Group 1 - Cohort 10 AMG 330 10/480 µg/Day | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day | Group 4 - Etanercept and AMG 330 | Group 4 - Etanercept, Dexamethasone and AMG 330 | Group 4: Tocilizumab, Dexamethasone and AMG 330
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 0/3 | 0/3 | 0/3 | 0/3 | 0/4 | 0/4 | 0/4 | 0/3 | 0/4 | 0/7 | 0/3 | 0/3 | 0/6 | 0/3 | 2/5 | 1/4 | 3/5 | 2/8 | 0/4 | 0/2 | 1/4 | 0/3 | 1/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/3 | 3/3 | 3/3 | 1/3 | 3/4 | 2/4 | 2/4 | 3/3 | 3/4 | 6/7 | 1/3 | 2/3 | 6/6 | 0/3 | 3/5 | 1/4 | 4/5 | 4/8 | 1/4 | 0/2 | 1/4 | 2/3 | 2/4 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 2/3 | 3/3 | 3/3 | 3/3 | 4/4 | 4/4 | 4/4 | 3/3 | 4/4 | 7/7 | 3/3 | 3/3 | 6/6 | 3/3 | 5/5 | 4/4 | 5/5 | 8/8 | 4/4 | 2/2 | 4/4 | 3/3 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Cohort 1 AMG 330 0.5 µg/Day (N=1) | Group 1 - Cohort 2 AMG 330 1.5 µg/Day (N=1) | Group 1 - Cohort 3 AMG 330 4 µg/Day (N=3) | Group 1 - Cohort 4 AMG 330 10 µg/Day (N=3) | Group 1 - Cohort 5 AMG 330 30 µg/Day (N=3) | Group 1 - Cohort 6 AMG 330 10/30 µg/Day (N=3) | Group 1 - Cohort 7 AMG 330 10/60 µg/Day (N=4) | Group 1 - Cohort 8 AMG 330 10/120 µg/Day (N=4) | Group 1 - Cohort 9 AMG 330 10/240 µg/Day (N=4) | Group 1 - Cohort 10 AMG 330 10/480 µg/Day (N=3) | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day (N=4) | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day (N=7) | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day (N=3) | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day (N=3) | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day (N=6) | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day (N=3) | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day (N=5) | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day (N=4) | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day (N=5) | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day (N=8) | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day (N=4) | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day (N=2) | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day (N=4) | Group 4 - Etanercept and AMG 330 (N=3) | Group 4 - Etanercept, Dexamethasone and AMG 330 (N=4) | Group 4: Tocilizumab, Dexamethasone and AMG 330 (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic neuropathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 3 | 1 | 0 | 1 | 2 | 2 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fournier's gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucormycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Cohort 1 AMG 330 0.5 µg/Day (N=1) | Group 1 - Cohort 2 AMG 330 1.5 µg/Day (N=1) | Group 1 - Cohort 3 AMG 330 4 µg/Day (N=3) | Group 1 - Cohort 4 AMG 330 10 µg/Day (N=3) | Group 1 - Cohort 5 AMG 330 30 µg/Day (N=3) | Group 1 - Cohort 6 AMG 330 10/30 µg/Day (N=3) | Group 1 - Cohort 7 AMG 330 10/60 µg/Day (N=4) | Group 1 - Cohort 8 AMG 330 10/120 µg/Day (N=4) | Group 1 - Cohort 9 AMG 330 10/240 µg/Day (N=4) | Group 1 - Cohort 10 AMG 330 10/480 µg/Day (N=3) | Group 1 - Cohort 11 AMG 330 10/60/240 µg/Day (N=4) | Group 1 - Cohort 12 AMG 330 10/60/240 ug/Day (N=7) | Group 1 - Cohort 13 AMG 330 10/60/360 µg/Day (N=3) | Group 1 - Cohort 14 AMG 330 10/60/480 µg/Day (N=3) | Group 1 - Cohort 15 AMG 330 10/240/600 µg/Day (N=6) | Group 1 - Cohort 16 AMG 330 10/240/600/720 µg/Day (N=3) | Group 1 - Cohort 17 AMG 330 10/240/600/840 µg/Day (N=5) | Group 1 - Cohort 18 AMG 330 10/240/600/960 µg/Day (N=4) | Group 1 - Cohort 19 AMG 330 10/240/600/960/1300 µg/Day (N=5) | Group 1 - Cohort 20 AMG 330 10/60/240/600/960/1600 µg/Day (N=8) | Group 2 - Cohort 1 AMG 300 30/240/600 µg/Day (N=4) | Group 2 - Cohort 2 AMG 330 30/240/840 µg/Day (N=2) | Group 3 - Cohort 1 AMG 330 30/240/600 µg/Day (N=4) | Group 4 - Etanercept and AMG 330 (N=3) | Group 4 - Etanercept, Dexamethasone and AMG 330 (N=4) | Group 4: Tocilizumab, Dexamethasone and AMG 330 (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 1 | 2 | 1 | 4 | 1 | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 1 | 3 | 3 | 4 | 1 | 0 | 4 | 2 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 1 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 3 | 1 | 1 | 5 | 2 | 0 | 2 | 3 | 4 | 2 | 1 | 3 | 1 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Intestinal dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 3 | 2 | 0 | 2 | 2 | 1 | 1 | 4 | 2 | 1 | 2 | 3 | 1 | 3 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 0 | 3 | 1 | 0 | 0 | 4 | 3 | 1 | 1 | 3 | 3 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 3 | 1 | 2 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema mucosal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 1 | 2 | 3 | 5 | 1 | 1 | 4 | 3 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 3 | 2 | 2 | 6 | 2 | 2 | 5 | 2 | 4 | 4 | 5 | 6 | 4 | 2 | 4 | 3 | 4 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoid infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes dermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia adenoviral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound decomposition (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ADAMTS13 activity decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Antithrombin III decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Antithrombin III increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Aspergillus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Blood bilirubin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 2 | 4 | 3 | 1 | 0 | 0 | 3 | 3 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT shortened (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunoglobulins increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interleukin level increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 2 | 2 | 1 | 0 | 3 | 2 | 0 | 0
Monocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 2 | 1 | 0 | 0
Procalcitonin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time shortened (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 0 | 2 | 3 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 4 | 2 | 0 | 0 | 4 | 3 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 2 | 1 | 0 | 2 | 3 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 3 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 2 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 2 | 0 | 1 | 1 | 4 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 3 | 1 | 2 | 3 | 2 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 2 | 3 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 3 | 1 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 2 | 1 | 3 | 2 | 2 | 3 | 3 | 1 | 1 | 2 | 3 | 2 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Protein deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 2 | 1 | 1 | 3 | 1 | 0 | 1 | 2 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 4 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonic clonic movements (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 2 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bruxism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depersonalisation/derealisation disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frustration tolerance decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocalyx (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Micturition frequency decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 2 | 2 | 3 | 1 | 1 | 0 | 1 | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 2 | 3 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 2 | 2 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 3 | 1 | 2 | 0 | 3 | 1 | 2 | 2 | 3 | 1 | 1 | 4 | 3 | 3 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 1 | 2 | 1 | 3 | 3 | 3 | 2 | 1 | 2 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 3 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 3 | 0 | 0 | 4 | 1 | 1 | 3 | 3 | 3 | 1 | 0 | 4 | 2 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5 | 1 | 1 | 3 | 2 | 0 | 2 | 2 | 3 | 0 | 1 | 1 | 2 | 2 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Group 5 dose-escalation cohort and dose-expansion cohorts were not enrolled in the study, due to the study terminating early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT02520427/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT02520427/SAP_001.pdf